CLINICAL TRIAL: NCT03554252
Title: Comparison of Different Frames of Numerical Information in Cochrane Plain Language: Randomized Controlled Trial
Brief Title: Comparison of Different Frames of Numerical Information in Cochrane Plain Language Summaries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 214-09-7672
Record Dates: First submitted 2018-05-17; First posted 2018-06-13 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-05

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frequencies (Experimental)
  Interventions: Other: Frequencies
- Percentages (Experimental)
  Interventions: Other: Percentages

INTERVENTIONS:
Other: Frequencies — Results are presented as natural frequencies (e.g. the drug was effective for 1 out of 10 people) while side effects are presented as percentages (e.g. 40% participants experienced severe side effects)
  Arms: Frequencies
Other: Percentages — Results are presented as percentages (e.g. the drug was effective for 10% of people) while side effects are presented as natural frequencies (e.g. 4 out of 10 participants experienced severe side effects)
  Arms: Percentages

SUMMARY:
Participants will be randomly given one of two formats containing descriptions of health interventions. In one format, participants will have to read short summaries where results of the intervention are presented as frequencies and the side effects of health intervention are presented as percentages, while in another format the frames will be reversed (results will be presented as percentages and side effects as frequencies). After reading, participants will be asked several questions about the content of the summary and its conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are visiting their family doctor, and are at least 18 old. Students of biomedical studies at University of Split School of Medicine, who are at least 18 years old.

Exclusion Criteria:

* Participants younger than 18 years.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Understanding | 3 months
  Number of the correct answers about the content of the summary, which will consist of four multiple choice questions (with four possible answers where only one is correct, for each question) about the text the participants are reading. Questions will be developed by research team and revised by expert in health communication. The scale ranges from 0-4, where greater score indicates better understanding of the material.

SECONDARY OUTCOMES:
Attitudes towards the appropriateness of this type of presentation of health information | 3 months
  Likert type scale from 1-10 (1 indicating low appropriateness and 10 would be completely appropriate presentation)
Health numeracy | 3 months
  5 questions about the numerical tasks placed in medical content, total score is number of correct answers on those questions. The five questions are part of Numeracy Understanding in Medicine Instrument (Schapira et al, 2012), and we will translate only the questions focusing on Probability section. Cronbach's alpha in previous research was 0.86 (Schapira et al, 2012). The questions will be revised by independent translator and back translated to English. The scale range is from 0-5, where higher score indicates higher numeracy levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Buljan, MPsy, Principal Investigator — PhD student
Locations (1):
- University of Split School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schapira MM, Walker CM, Cappaert KJ, Ganschow PS, Fletcher KE, McGinley EL, Del Pozo S, Schauer C, Tarima S, Jacobs EA. The numeracy understanding in medicine instrument: a measure of health numeracy developed using item response theory. Med Decis Making. 2012 Nov-Dec;32(6):851-65. doi: 10.1177/0272989X12447239. Epub 2012 May 25. PMID 22635285
- [Derived] Buljan I, Tokalic R, Roguljic M, Zakarija-Grkovic I, Vrdoljak D, Milic P, Puljak L, Marusic A. Framing the numerical findings of Cochrane plain language summaries: two randomized controlled trials. BMC Med Res Methodol. 2020 May 6;20(1):101. doi: 10.1186/s12874-020-00990-4. PMID 32375659